CLINICAL TRIAL: NCT04347590
Title: Impact of Continuous Glucose Monitoring on Cerebral Oxygenation in Preterm Infants (the Babyglucolight Trial)
Brief Title: Continuous Glucose Monitoring and Cerebral Oxygenation in Preterm Infants
Acronym: Glucolight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Alfonso Galderisi, MD, PhD, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AOP1813
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Infant Development; Hypoglycemia Neonatal; Neurodevelopmental Abnormality
Keywords: continuous glucose monitoring (cgm); neonatal hypoglycemia; preterm infants; diffuse optical tomography (dot)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Unblinded CGM (Experimental): CGM data will be "unblinded", with Hypo/hyperglycemia alarms on. Data will be recorded from CGM every three hours and intervention to adequate glucose intake will be performed to keep glycemia in normal range (72-144mg/dl) if necessary.
  Interventions: Device: Unblinded - CGM (Medtronic Guardian)
- Blinded CGM (Other): Hypo/hyper alarms are off. CGM data will be blinded. Glucose intake will be adequate according to at least 2 capillary glycemic tests per day.
  Interventions: Device: Blinded - CGM (Medtronic Guardian)

INTERVENTIONS:
Device: Unblinded - CGM (Medtronic Guardian) — Data from device will be readable and alarms on
  Arms: Unblinded CGM
Device: Blinded - CGM (Medtronic Guardian) — Data from device will be blinded and alarms off
  Arms: Blinded CGM

SUMMARY:
Neonatal hypoglicaemia is associated with impaired neurodevelopment outcomes in preterm infants. Thus, hypoglicemic events should be diagnosed and treated promptly. Unfortunately, hypo- and hyperglicaemia management is still controversial.

The investigators aim to assess if a continuous glucose monitor (CGM) impacts on both short-term and long-term neurodevelopment. Primary outcome is the effect of CGM coupled with a control algorithm for glucose infusion on the number of hemodynamic significant events (defined as hypoglycemic events associated with DOT-detectable reduction of brain oxygenation).

It will be enrolled newborns ≤32 weeks gestational age and/or of birthweight ≤1500 g, they will be randomized in two study arms, both of them will wear Medtronic CGM during the first 5 days of life: 1) Blinded group (B): the device monitor will be switched off, glucose infusion rate will be modified according to the daily capillary glucose tests. 2) Unblinded group (UB): the device monitor will be visibile, alarms for hypos/hyper will be active and glucose infusion rate will be modulated according to CGM and PID control algorithm.

Enrolled newborns will also be monitored with near-infrared diffuse optical tomography (DOT) during the first 5 days from enrollment.

Follow-up will be performed at 12, 18, 24 months and 5 years by neurodevleopmental scale (Bailey III until 24 months; Wechsler Preschool and Primary Scale of Intelligence (WPPSI) at 5 years).

The estimated numerosity is 60 patients (30 for each arm).

DETAILED DESCRIPTION:
Background - Hypoglycaemia is a very common event during the first week of life, it affects up to 15% of term newborns and it is more frequent in preterm and IUGR (Intrauterine Growth Restriction with birth weight <10th percentile) infants.

Repeated and prolonged hypoglicemic events are associated with impaired neurodevelopment outcomes in preterm infants and should be diagnosed and treated promptly (Tam EWY et al, J Pediatrics 2012; Duvanel et al, J Ped 1999; Lucas et al BMJ; 1988; Filam PM et al, J Pediatr 2006).

Unfortunately, the management of hypo / hyperglycaemias in these groups is still controversial due to the lack of Continuous Glucose Monitoring System's (CGMS) efficacy assessments in the Neonatal Care Intensive Units.

Nevertheless, recent studies indicate that CGMS is reliable and can identify a significant number of hypoglycaemias (<40mg / dl, duration> 30 minutes) which could not be recognized through traditional glycemic monitoring (Pertierra Cortada et al, J Ped 2014; Beardsall et al, Arch Dis Child Fetal&Neonatal Ed 2013).

The reliability of data provided by CGMS were highlighted by Beardsall and colleagues (Beardsall et al, Arch Dis Child Fetal & Neonatal Ed 2013) on a population of newborns with an average birth weight of 1007 gr (SD 0.27) and a gestational age of 28.36 SG (SD 2.26), the study showed a high correlation (0.94) between capillary monitoring data (traditional) and data provided by the CGMS.

However, the effects of these CGMS-based approaches on short and long-term neurodevelopment are still unknown, as well as the real impact of these glycemic variations and the maintenance of euglycemia on cerebral hemodynamics.

Indeed, every treatment proposed in this fragile population must have, as its ultimate aim, the improvement of its neuro-cognitive development in order to be considered effective and useful.

Aim - The study the Investigators are going to conduct is aimed to evaluate if CGM, as driver of therapeutic decisions in preterm newborns (birthweight ≤1500g, gestational age ≤32 weeks) during the first week of life, may be able to improve both short-term and long-term neurodevelopment.

Study design - Randomized Controlled Trial

* Patients: newborns with GA ≤32weeks and/or BW≤ 1500 g. They will be enrolled within the first 48 hours of life
* Intervention group: Unblinded CGM + Proportional integrative Derivative algorithm (PID) to adequate daily glucose intake
* Control group: Blinded CGM with daily glucose intake adequated according to SMBG (=2 blood glucose/day) using standard of care (ESPGHAN) intakes
* Primary Outcome: to evaluate if the use of CGMS (Continuous glucose monitoring system) combined with an algorithm for glucose infusion reduces the number of hemodynamically significant hypoglycemic events during the first week of life

Matherials and Methods - Continuous glucose sensor (Medtronic guardian) will be applied within 48 hours from birth to the study population on the lateral side of thigh, after parents' consent collection.

All the patients will be randomized to the blinded or unblinded group before the application of CGM. Randomization will be performed using a randomization list electronically generated.

Near-infrared diffuse optical tomography (DOT) will be used for brain monitoring. The instrumentation consists of:

* A cap, similar to the one we already created and used in a pilot study in this population (Galderisi et al., Neurophotonics 2016)
* Optical fibers, connected to the instrumentation and inserted into specific holes for optodes placed in the cap
* An external device containing lasers and detectors, controlled by a portable personal computer

Blinded group: they will wear CGM for 5 days, the alarms and the CGM monitor will be switched off. The daily amount of carbohydrates will be decided according to blood glucose tests (at least 2 per day).

Unblinded group (intervention/open CGM group): they will wear CGM for 5 days, the alarms of CGM will be switched on. The daily intake of carbohydrates will be adapted according to CGM data. In case of reported hypoglicaemia (<47 mg/dl), the data will be confirmed by capillary / catheter blood sampling and it wil be treated with Dextrose 40% gel (200 mg/kg) or 2 mg/kg 10% glucose solution.

Glucose adjustment for values out of the target tight glycemic range (72-144mg/dL) will be decided according to the PID algorithm and performed every 3 hours as suggested by the algorithm.

Numerosity: the estimated numerosity is 60 patients. (30 per arm)

Reasons for study interruption: local and/or systemic complication due to the application of device, transfer of patient to another center of care, withdrawal of consent, death, malfunction of device. Reasons for interruption of monitoring will be specified in the final report.

Risks and benefits analysis - The open CGM is expected to decrease the duration and number of hypoglicemic episodes. Early detection of the hypoglicemic events helps reducing their frequency, while adaptation of carbohydrate intake based on CGM data will prevent further hypoglycemic episodes during the observation period.

In addition, this device permits to reduce the number of blood sampling in the U-CGM group, reducing a painful (heel stick) and potentially dangerous (catheter sampling) procedure.

Even though the risk of local reaction is conceivable, it has never been described in studies conducted in newborns. If a local reaction occurs, the device will be removed and the trial will end for the patient.

Perspective and limits - Although the use of the CGMS in preterm infants has been well described, its efficacy in improving short-term and long-term neurodevelopment has never been established, as well as the connection between glycaemic variations and cerebral activity in this population. Only by achieving this goal the real efficacy and utility of CGMS in this population will be clear.

The study has been designed as a no-profit research project by the Principal Investigators and Collaborators of Neonatal Intensive Care Unit of University of Padua.

Interim assessment: after 20 participants enrolled; subsequent interim assessment have been planned every 20 participants enrolled. Study will be interrupted if >10% difference in primary outcome.

Funding: STARS grant from University of Padova (Italy); Penta Foundation; CARIPARO

ELIGIBILITY:
Inclusion Criteria:

* <= 32 weeks gestation
* birthweight <1500 g

Exclusion Criteria:

* birthweight <500g
* congenital pathologies
* lack of parental consent
* perinatal maternal infections
* albinism

Ages: 2 Hours to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
CGMS and brain hemodynamic (posterior areas) | 5 days
  Number of hypoglycemic events henomdynamically significant. Hypoglycemic events are defined as any value <72mg/dL (mild hypo) or <47mg/dL (severe hypo). They are classified as "significant" in the presence of a reduction from baseline HbT >=15% (posterior areas)

SECONDARY OUTCOMES:
CGMS and brain hemodynamic (overall) | 5 days
  Number of hypoglycemic events henomdynamically significant. Hypoglycemic events are defined as any value <72mg/dL (mild hypo) or <47mg/dL (severe hypo). They are classified as "significant" in the presence of a reduction from baseline HbT >=15% (average of tested areas)
Long-term neurodevelopment | 24 months
  Effect of CGM based intervention on Bayley III performance at 24 months
Long-term neurodevelopment 2 | 12 months
  Effect of CGM based intervention on Bayley III performance at 12 months
Long-term neurodevelopment 3 | 18 months
  Long-term neurodevelopment on Bayley III performance at 18 months
Long-term neurodevelopment 4 | 36 months
  Long-term neurodevelopment on Bayley III performance at 36 months
Long-term neurodevelopment 4 | 50 months
  Long-term neurodevelopment on Bayley III performance at 50 months
CGMS and brain hemodynamic (overall-hyperglycemia) | 5 days
  Effect of Hyperglycemia (>144mg/dL and >180mg/dL) on brain hemodynamic
Intervention and brain hemodynamic | 5 days
  effect of intervention on overall brain hemodynamic (baseline vs end of study monitoring DOT)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Galderisi, MD, Principal Investigator — University Hospital of Padua
Locations (1):
- Neonatal Intensive Care Unit - University Hospital of Padua, Padua, Italy

REFERENCES:
- [Result] Agus MS, Steil GM, Wypij D, Costello JM, Laussen PC, Langer M, Alexander JL, Scoppettuolo LA, Pigula FA, Charpie JR, Ohye RG, Gaies MG; SPECS Study Investigators. Tight glycemic control versus standard care after pediatric cardiac surgery. N Engl J Med. 2012 Sep 27;367(13):1208-19. doi: 10.1056/NEJMoa1206044. Epub 2012 Sep 7. PMID 22957521
- [Result] Beardsall K, Vanhaesebrouck S, Ogilvy-Stuart AL, Vanhole C, VanWeissenbruch M, Midgley P, Thio M, Cornette L, Ossuetta I, Palmer CR, Iglesias I, de Jong M, Gill B, de Zegher F, Dunger DB. Validation of the continuous glucose monitoring sensor in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2013 Mar;98(2):F136-40. doi: 10.1136/archdischild-2012-301661. Epub 2012 Jul 12. PMID 22791467
- [Result] Beardsall K, Vanhaesebrouck S, Ogilvy-Stuart AL, Vanhole C, Palmer CR, van Weissenbruch M, Midgley P, Thompson M, Thio M, Cornette L, Ossuetta I, Iglesias I, Theyskens C, de Jong M, Ahluwalia JS, de Zegher F, Dunger DB. Early insulin therapy in very-low-birth-weight infants. N Engl J Med. 2008 Oct 30;359(18):1873-84. doi: 10.1056/NEJMoa0803725. PMID 18971490
- [Result] Chalia M, Lee CW, Dempsey LA, Edwards AD, Singh H, Michell AW, Everdell NL, Hill RW, Hebden JC, Austin T, Cooper RJ. Hemodynamic response to burst-suppressed and discontinuous electroencephalography activity in infants with hypoxic ischemic encephalopathy. Neurophotonics. 2016 Jul;3(3):031408. doi: 10.1117/1.NPh.3.3.031408. Epub 2016 May 2. PMID 27446969
- [Result] Debillon T, Zupan V, Ravault N, Magny JF, Dehan M. Development and initial validation of the EDIN scale, a new tool for assessing prolonged pain in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2001 Jul;85(1):F36-41. doi: 10.1136/fn.85.1.f36. PMID 11420320
- [Result] Russell SJ, El-Khatib FH, Sinha M, Magyar KL, McKeon K, Goergen LG, Balliro C, Hillard MA, Nathan DM, Damiano ER. Outpatient glycemic control with a bionic pancreas in type 1 diabetes. N Engl J Med. 2014 Jul 24;371(4):313-325. doi: 10.1056/NEJMoa1314474. Epub 2014 Jun 15. PMID 24931572
- [Result] Shah VS, Ohlsson A. Venepuncture versus heel lance for blood sampling in term neonates. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD001452. doi: 10.1002/14651858.CD001452.pub4. PMID 21975734
- [Result] Sinclair JC, Bottino M, Cowett RM. Interventions for prevention of neonatal hyperglycemia in very low birth weight infants. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD007615. doi: 10.1002/14651858.CD007615.pub3. PMID 21975772
- [Result] Singh H, Cooper RJ, Wai Lee C, Dempsey L, Edwards A, Brigadoi S, Airantzis D, Everdell N, Michell A, Holder D, Hebden JC, Austin T. Mapping cortical haemodynamics during neonatal seizures using diffuse optical tomography: a case study. Neuroimage Clin. 2014 Jul 6;5:256-65. doi: 10.1016/j.nicl.2014.06.012. eCollection 2014. PMID 25161892
- [Result] Duvanel CB, Fawer CL, Cotting J, Hohlfeld P, Matthieu JM. Long-term effects of neonatal hypoglycemia on brain growth and psychomotor development in small-for-gestational-age preterm infants. J Pediatr. 1999 Apr;134(4):492-8. doi: 10.1016/s0022-3476(99)70209-x. PMID 10190926
- [Result] Filan PM, Inder TE, Cameron FJ, Kean MJ, Hunt RW. Neonatal hypoglycemia and occipital cerebral injury. J Pediatr. 2006 Apr;148(4):552-5. doi: 10.1016/j.jpeds.2005.11.015. PMID 16647423
- [Result] Galderisi A, Brigadoi S, Cutini S, Moro SB, Lolli E, Meconi F, Benavides-Varela S, Baraldi E, Amodio P, Cobelli C, Trevisanuto D, Dell'Acqua R. Long-term continuous monitoring of the preterm brain with diffuse optical tomography and electroencephalography: a technical note on cap manufacturing. Neurophotonics. 2016 Oct;3(4):045009. doi: 10.1117/1.NPh.3.4.045009. Epub 2016 Dec 23. PMID 28042587
- [Result] Mitanchez D. Glucose regulation in preterm newborn infants. Horm Res. 2007;68(6):265-71. doi: 10.1159/000104174. Epub 2007 Jun 20. PMID 17587854
- [Result] Harris DL, Battin MR, Weston PJ, Harding JE. Continuous glucose monitoring in newborn babies at risk of hypoglycemia. J Pediatr. 2010 Aug;157(2):198-202.e1. doi: 10.1016/j.jpeds.2010.02.003. Epub 2010 Mar 24. PMID 20338573
- [Result] Hay WW Jr, Raju TN, Higgins RD, Kalhan SC, Devaskar SU. Knowledge gaps and research needs for understanding and treating neonatal hypoglycemia: workshop report from Eunice Kennedy Shriver National Institute of Child Health and Human Development. J Pediatr. 2009 Nov;155(5):612-7. doi: 10.1016/j.jpeds.2009.06.044. No abstract available. PMID 19840614
- [Result] Rozance PJ, Hay WW. Hypoglycemia in newborn infants: Features associated with adverse outcomes. Biol Neonate. 2006;90(2):74-86. doi: 10.1159/000091948. Epub 2006 Mar 9. PMID 16534190
- [Result] Lucas A, Morley R, Cole TJ. Adverse neurodevelopmental outcome of moderate neonatal hypoglycaemia. BMJ. 1988 Nov 19;297(6659):1304-8. doi: 10.1136/bmj.297.6659.1304. PMID 2462455
- [Result] Mena P, Llanos A, Uauy R. Insulin homeostasis in the extremely low birth weight infant. Semin Perinatol. 2001 Dec;25(6):436-46. doi: 10.1053/sper.2001.30349. PMID 11778914
- [Result] Pertierra-Cortada A, Ramon-Krauel M, Iriondo-Sanz M, Iglesias-Platas I. Instability of glucose values in very preterm babies at term postmenstrual age. J Pediatr. 2014 Dec;165(6):1146-1153.e2. doi: 10.1016/j.jpeds.2014.08.029. Epub 2014 Sep 24. PMID 25260622
- [Result] Iglesias Platas I, Thio Lluch M, Pociello Alminana N, Morillo Palomo A, Iriondo Sanz M, Krauel Vidal X. Continuous glucose monitoring in infants of very low birth weight. Neonatology. 2009;95(3):217-23. doi: 10.1159/000165980. Epub 2008 Oct 30. PMID 18971588
- [Result] Staffler A, Klemme M, Mola-Schenzle E, Mittal R, Schulze A, Flemmer AW. Very low birth weight preterm infants are at risk for hypoglycemia once on total enteral nutrition. J Matern Fetal Neonatal Med. 2013 Sep;26(13):1337-41. doi: 10.3109/14767058.2013.784250. Epub 2013 Apr 17. PMID 23528249
- [Result] Tam EW, Haeusslein LA, Bonifacio SL, Glass HC, Rogers EE, Jeremy RJ, Barkovich AJ, Ferriero DM. Hypoglycemia is associated with increased risk for brain injury and adverse neurodevelopmental outcome in neonates at risk for encephalopathy. J Pediatr. 2012 Jul;161(1):88-93. doi: 10.1016/j.jpeds.2011.12.047. Epub 2012 Feb 4. PMID 22306045
- [Result] Tin W, Brunskill G, Kelly T, Fritz S. 15-year follow-up of recurrent "hypoglycemia" in preterm infants. Pediatrics. 2012 Dec;130(6):e1497-503. doi: 10.1542/peds.2012-0776. Epub 2012 Nov 5. PMID 23129080
- [Result] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730